CLINICAL TRIAL: NCT05722704
Title: Effect of Cryotherapy and Occlusal Reduction on Post-endodontic Pain in Patients With Symptomatic Apical Periodontitis
Brief Title: Effect of Cryotherapy on Post-endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Principal Investigator, Rania Zaarour, Assistant Professor of Cell Biology and Researcher, Gulf Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB/COD/STD/14/May-2022
Record Dates: First submitted 2023-01-23; First posted 2023-02-10 (Actual); Results first posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-11

CONDITIONS: Cryotherapy
Keywords: Post endodontic pain; Cryotherapy; Occlusal reduction; Root canal treatment
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cryotherapy (Experimental): Final irrigation with cold saline (2.5C-4C) without occlusal reduction
  Interventions: Procedure: Cryotherapy
- Occlusal reduction (Active Comparator): Normal room temperature saline irrigation protocol with occlusal reduction
  Interventions: Procedure: Occlusal reduction
- Control (No Intervention): Normal room temperature saline irrigation protocol without occlusal reduction

INTERVENTIONS:
Procedure: Cryotherapy — Final irrigation with cold saline (2.5C-4C) without occlusal reduction
  Arms: Cryotherapy
Procedure: Occlusal reduction — Reduction of the functional and non-functional cusps
  Arms: Occlusal reduction

SUMMARY:
The goal of this clinical trial is to compare Cryotherapy with occlusal reduction in the reduction of post-endodontic pain in molars with symptomatic apical periodontitis. The main question it aims to answer is:

Is there is a difference in post-endodontic pain intensity following cryotherapy or occlusal reduction in patients with symptomatic apical periodontitis on mandibular first molars?

Participants will undergo root canal treatment including cryotherapy or post-operative occlusal reduction.

Researchers will compare [Cryotherapy, occlusal reduction, and no intervention] to see the intensity of post-endodontic pain.

DETAILED DESCRIPTION:
The study will be conducted on 60 first mandibular molars; with 20 first mandibular molars in each group (n=20). The patient will be asked to pick an opaque sealed envelope that will contain a number from 1 to 3. The resultant number will determine in which group the participants will be placed. Double blinding will be maintained in this study as the operator and the patients will not be aware of their group/used root canal irrigant.

Group I : normal room temperature saline irrigation protocol without occlusal reduction.

Group II : normal room temperature saline irrigation protocol with occlusal reduction.

Group III : final irrigation with cold saline (2.5 C°- 4 C°) without occlusal reduction.

Procedural steps:

1. Vitality will be assessed using cold tests and electric pulp testing before the procedure is carried out. Besides, mobility, palpation, and percussion tests will be done to assess periapical health. In order to ensure that the cold and electrical pulp tests are working, and a response is elicited, both tests will be carried out on patients not included in the study.
2. All the patients will receive local anesthesia: 2% lidocaine with 1:100,000 epinephrine.
3. Each tooth will be isolated using a rubber dam, and the access cavity will be prepared using a round bur (no.4) and tapered fissure diamond bur under copious water.
4. After removal of coronal pulp tissues using a sterile excavator, the working length will be determined with stainless steel hand K-files size #10 and the use of an apex locator and confirmed using intraoral periapical radiographs.
5. Hand instrumentation to 15-size K files.
6. All the canals will be prepared using ProTaper Gold rotary files till the master apical file F2.
7. Apical patency will be maintained throughout the shaping procedure using the #10 file between each instrument.
8. All the canals will be irrigated with 10 mL of 3% NaOCl between each file during the whole preparation procedure.
9. In group I the root canals will be obturated directly after preparation.
10. In group II occlusal reduction will be performed after root canal preparation.
11. For group III the root canals will be irrigated for 5 min using 20 ml cryo-treated saline maintained at a temperature of 2°C-4°C.
12. After completion of cleaning and shaping dried using appropriate size paper points and the canals will be obturated using gutta-percha, and restored by permanent composite restoration.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-70 years
2. A patient diagnosed with symptomatic irreversible pulpitis/acute apical periodontitis
3. require endodontic therapy
4. Mandibular first molars that are diagnosed with symptomatic irreversible pulpitis/acute apical periodontitis
5. Healthy patients without systemic disease
6. Permanent mature first mandibular molars

Exclusion Criteria:

1. Medically compromised patients
2. Pregnant patients
3. Teeth with incomplete apex formation
4. Teeth with calcified canals
5. Periapical abscess
6. Patients on antibiotic therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-12-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf Medical University, Ajman, United Arab Emirates

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cryotherapy | Occlusal Reduction | Control
Started | 20 | 20 | 20
Completed | 20 | 20 | 20
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cryotherapy | Occlusal Reduction | Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (7.85) | 31.4 (6.56) | 32.35 (8.98) | 32.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 17 | 12 | 40
  Male | 9 | 3 | 8 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 20 | 20 | 20 | 60
Region of Enrollment [Count of Participants; unit: Participants]
  United Arab Emirates | 20 | 20 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: The Level of Post-endodontic Pain
Description: Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be)
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Occlusal Reduction: Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be
- Saline: Evaluation of the pain intensity using the Visual Analogue Scale. The Visual Analogue Scale measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two endpoints representing 0 ('no pain') and 10 ('pain as bad as it could possibly be)
Arm/Group | Cryotherapy | Occlusal Reduction | Saline
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 1.85 (1.81) | 2.15 (2.11) | 3.65 (3.03)
Statistical Analysis 1: Comparison: Cryotherapy vs Occlusal Reduction; Test type: Superiority; p = 0.986, Kruskal-Wallis; Median Difference (Net) = 0.118, Standard Deviation 0.05

2. Primary Outcome: The Level of Post-endodontic Pain
Description: as for outcome 1
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryotherapy | Occlusal Reduction | Saline
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.70 (1.13) | 1.2 (1.32) | 2.2 (1.82)
Statistical Analysis 1: Comparison: Cryotherapy vs Occlusal Reduction; Test type: Superiority; p < 0.118, Kruskal-Wallis; Median Difference (Net) = 0.016, Standard Deviation 0.05

3. Primary Outcome: The Level of Post-endodontic Pain
Description: as for outcome 1
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cryotherapy | Occlusal Reduction | Saline
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.25 (0.79) | 1.2 (1.32) | 2.2 (1.82)
Statistical Analysis 1: Comparison: Cryotherapy vs Occlusal Reduction; Test type: Superiority; p = 0.225, Kruskal-Wallis; Median Difference (Net) = 95, Standard Deviation 0.05

4. Primary Outcome: The Level of Post-endodontic Pain
Description: as for outcome 1
Time Frame: 72 hours
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Cryotherapy | Occlusal Reduction | Saline
Number analyzed (Participants) | 20 | 20 | 20
score on a scale | 0.10 (0.45) | 0.05 (0.22) | 0.25 (0.72)
Statistical Analysis 1: Comparison: Cryotherapy vs Occlusal Reduction; Test type: Superiority; p = 0.424, Kruskal-Wallis; Median Difference (Net) = 95, Standard Deviation 0.05

ADVERSE EVENTS:
Time Frame: at 3 month, 6 month, and 1 year.
Description: Overall number of participants, in each arm/group, who died due to any cause.
Groups:
- Saline: Normal room temperature saline irrigation protocol without occlusal reduction
Arm/Group | Cryotherapy | Occlusal Reduction | Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT05722704/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2024-11-13): https://cdn.clinicaltrials.gov/large-docs/04/NCT05722704/SAP_001.pdf